CLINICAL TRIAL: NCT05370118
Title: Improving Physical Activity With Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2002895
Record Dates: First submitted 2022-03-15; First posted 2022-05-11 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Mild Cognitive Impairment; Caregiver Burnout
Keywords: physical activity; behavior change
MeSH Terms: conditions — Cognitive Dysfunction; Caregiver Burden; Motor Activity | interventions — Methods

STUDY DESIGN:
Intervention Model Description: This pilot clinical research study is structured as a feasibility and preliminary efficacy trial to determine if the TPAB intervention is feasible and to compare daily step improvement between the TPAB intervention group and the CTL group. The trial is designed to inform a future larger-scale efficacy trial to assess longer time points for the sustainability of intervention impact.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors will be masked from the participant's treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation physical activity behavioral (TPAB) intervention (Experimental): Individuals in the TPAB intervention will participate in a weekly session for 12 weeks with their primary caregiver and the research interventionist (RH). Established behavior-change techniques will be used in the TPAB intervention, based largely on the combination of the Social Cognitive Theory, Control Theory, and Operant Conditioning,43 including behavioral techniques, and patient-centered communication (e.g., motivational interviewing).44 The behavior-change techniques are designed to target and improve daily steps. Individuals in the CTL group will receive usual care and no intervention over the 12 weeks.
  Interventions: Behavioral: Telerehabilitation physical activity behavioral (TPAB) intervention
- Control Group (No Intervention): Individuals in the CTL group will receive usual care and no intervention over the 12 weeks.

INTERVENTIONS:
Behavioral: Telerehabilitation physical activity behavioral (TPAB) intervention — The intervention includes the behavior change techniques of self-monitoring of behavior, action planning, graded tasks, restructuring the physical and social environment, problem-solving, and prompts/cues.
  Arms: Telerehabilitation physical activity behavioral (TPAB) intervention

SUMMARY:
Individuals with mild cognitive impairment are often physically inactive and at risk for progressing to dementia. Physical inactivity is considered a modifiable risk factor for dementia. Therefore, interventions must be developed to foster sustainable improvement in daily physical activity. To address this problem, our pilot study aims are directed at assessing the feasibility and preliminary improvement of physical activity following the use of a mobile-health technology physical activity behavior change intervention. Similar interventions have shown to be very effective in older adults without cognitive impairment. We specifically focus on the subtype of amnestic mild cognitive impairment since this subtype often progresses to Alzheimer's Disease, a leading cause of death in the US. Improving physical activity is one approach to reduce the progression to Alzheimer's Disease and subsequently lower mortality. To increase the impact of the intervention, participants with amnestic mild cognitive impairment will be recruited along with a primary caregiver (dyads). Thirty dyads will be recruited and randomized to either an intervention group (15 dyads) or usual care group (15 dyads). The intervention group will receive a 12-week mobile-health technology physical activity behavior change intervention structured to improve physical activity. The intervention is unique in the combination of established behavior change theories and techniques and remote delivery for individuals with amnestic mild cognitive impairment. This pilot study is designed to assess the feasibility of the intervention by examining participant and primary caregiver retention, intervention session attendance, intervention acceptability and safety, and qualitative perspectives. Secondly, this pilot study will assess preliminary improvement in physical activity (i.e., daily steps). Improvement will be determined based on significant changes in participants' daily steps observed via accelerometry post-intervention in the intervention group compared to the usual care control group. The results of this study will support future work (K-award and R01 submissions) to explore efficacy and larger-scale implementation to reach rural and underserved areas of Nebraska and beyond.

DETAILED DESCRIPTION:
The primary objective of this pilot study is to determine the feasibility and preliminary efficacy of a telerehabilitation physical activity behavioral (TPAB) intervention for improving habitual physical activity in individuals with amnestic mild cognitive impairment (MCI).

Amnestic MCI is considered a precursor to Alzheimer's Disease (AD), the sixth leading cause of death in the US.1 Additionally, loss of independence and cognitive function is one of the most feared aspects of aging for older adults.2,3 One way to promote independence is through physical activity. Physical inactivity is highly reported in those with MCI4 and is a modifiable risk factor for those with dementia.5,6 Therefore, strategies to combat the loss of physical independence and cognition are of high economic and quality of life priority.

Home-based physical activity behavior change methods have successfully improved physical activity in healthy older adults7-10 but have had limited use in individuals with MCI.11 This study will determine the feasibility and preliminary efficacy of the TPAB intervention in individuals with amnestic MCI and caregivers to provide the groundwork to ascertain clinical implementation. In this randomized controlled clinical research study, we will assess the feasibility and preliminary efficacy of the TPAB intervention in individuals with amnestic MCI. The TPAB intervention consists of 12 telerehabilitation sessions (30 min) over 12 weeks. Primary caregivers will be included during all intervention sessions based on dyadic approaches demonstrating higher physical activity invention success in individuals with MCI compared to individual recruitment.12 The TPAB intervention group will include 15 dyads of patients with amnestic MCI and their primary caregivers. The TPAB intervention is an evidence-based intervention designed to improve daily steps in older adults with medical complexities.13-15 It combines strategies such as problem-solving11, action planning16, and motivational interviewing17 that are evidenced to improve physical activity in individuals with MCI.11,16,17 The TPAB intervention will require a wearable sensor (Fitbit) and a home-based tablet/laptop to allow real-time activity feedback and video interface between participants and the interventionist. The TPAB intervention is novel in combining theories and techniques and remote delivery for individuals with amnestic MCI. The control (CTL) group will include 15 dyads of individuals with amnestic MCI and their primary caregivers that will receive usual care over the 12 weeks. Outcomes for both groups will be assessed before the intervention (baseline) and at the end of the intervention (POST). The specific aims are:

Aim 1: Determine the feasibility of the TPAB intervention for individuals with amnestic MCI and their primary caregivers by measuring 1) participant retention, 2) attendance, 3) acceptability (Intrinsic Motivation Inventory18), 3) safety (adverse event tracking), 4) semi-structured interviews.

Aim 2: Examine the preliminary effects of TPAB on physical activity engagement among MCI participants when compared with the CTL group.

Hypothesis 2.1: Individuals with amnestic MCI will make significant (p<0.05) gains in accelerometer-assessed (activPAL) physical activity (daily steps) from baseline to POST compared to the CTL group.

Clinical Impact: This study addresses two significant clinical gaps for amnestic MCI rehabilitation: 1) lack of evidence-based rehabilitation strategies to improve habitual physical activity; and 2) barriers to remotely promote habitual physical activity. Lastly, this project will bring together an interdisciplinary team (physical therapist (RH), exercise scientist (DE), and neuropsychologist (VP)) of investigators at Creighton University and the University of Nebraska Medical Center (UNMC).

ELIGIBILITY:
Inclusion Criteria:

1. 50-85 years old (patient); 19+ years (caregiver)
2. clinically diagnosed with amnestic MCI (patient only)
3. a score of 18-24 on the Montreal Cognitive Assessment indicating possible MCI (patient only),
4. not currently categorized as "Active" on the Rapid Assessment of Physical Activity, (patient only)
5. on stable doses of medication at least for the previous 30 days at baseline (patient only)
6. have a computer/wireless device with Internet access
7. have a primary caregiver willing to participate in physical activity and assist the patient with participation in the study
8. English-speaking

Exclusion Criteria:

1. limitations due to disability, illness, or pain that may affect the patient's walking safety during the study
2. unstable heart conditions (e.g., unstable angina, acute pericarditis)
3. uncontrolled hypertension in the last six months
4. known neurological diseases

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
TPAB intervention Participant Retention | The outcome will be reported at the end of the 12 week intervention.
  The number of participants that complete the 12 week intervention will be calculated to determine participant retention.
TPAB Intervention Attendance | The outcome will be reported at the end of the 12 week intervention.
  The number of weekly sessions attended across the 12-week intervention will be totaled to determine the TPAB Intervention Attendance.
TPAB Intervention Acceptability | The outcome will be reported at the end of the 12 week intervention.
  The acceptability of the TPAB Intervention will be assessed by administering the Intrinsic Motivation Inventory Interest/Enjoyment Subscale at the conclusion of the intervention. The Intrinsic Motivation Inventory Subscale includes 7 statements that require the participant to respond on a 1-7 scale to the level they agree with the statement. The total score ranges from 7-49 with higher scores indicating greater Interest/Enjoyment.
TPAB Intervention Safety | The outcome will be reported at the end of the 12 week intervention.
  The safety of the TPAB Intervention will be assessed by tracking and comparing the number of adverse events in the intervention and control group.
Feasibility of the TPAB Intervention (Semi-Structured Interviews) | Semi-Structured Interviews will be conducted at the end of the 12 week intervention.
  Semi-structured interview will be conducted on the patient and caregivers that participated in the TPAB Intervention. Qualitative analysis will determine common themes in the responses.

SECONDARY OUTCOMES:
Daily step count change | Baseline and after the 12 week intervention
  daily step count will be measured with the activPAL physical activity monitor over a seven day period

CONTACTS AND LOCATIONS:
Locations (1):
- Creighton University, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data will be available upon request. Other data sharing is undecided at this time.